CLINICAL TRIAL: NCT03236649
Title: Comparison of Efficacy and Safety of Icaritin Versus Sorafenib in First-line Treatment of PD-L1 Positive Advanced Hepatocellular Carcinoma Subjects: a Multicenter, Randomized, Opened Phase III Clinical Trial
Brief Title: The Phase III Study of Icaritin Versus Sorafenib in PD-L1 Positive Advanced Hepatocellular Carcinoma Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Because the clinical development plan has been changed.
Sponsor: Beijing Shenogen Biomedical Co., Ltd (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Eastern Theater General Hospital,QinHuai District Medical Area (Unknown); Peking University Cancer Hospital & Institute (Other); Chinese PLA General Hospital (Other); Beijing Hospital (Other Government); General Hospital of Chinese Armed Police Forces (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Jinan Central Hospital (Other); Linyi Cancer Hospital (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Anhui Provincial Hospital (Other Government); The First Affiliated Hospital with Nanjing Medical University (Other); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); Nanfang Hospital, Southern Medical University (Other); First People's Hospital of Foshan (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Hebei Medical University Fourth Hospital (Other); Hunan Cancer Hospital (Other); The First Hospital of Jilin University (Other); 307 Hospital of PLA (Other); Fudan University (Other); Henan Cancer Hospital (Other Government); Jilin Provincial Tumor Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital of Bengbu Medical University (Other); The First Affiliated Hospital of Soochow University (Other); Tongji Hospital (Other); Beijing YouAn Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNG1705ICR-2
Record Dates: First submitted 2017-07-26; First posted 2017-08-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2021-01

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — icaritin; Sorafenib

STUDY DESIGN:
Intervention Model Description: Open, randomized controlled, multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Icaritin (Experimental): 600mg/time, 6 capsules/time(6×100mg/capsule), 2 times/day(30 minutes after breakfast, lunch and dinner), take orally, continuous administration until reach the standard of termination.
  Interventions: Drug: Icaritin
- Sorafenib Tosylate Tablets (Active Comparator): 400mg/time, 2 tablets/time(2×200mg/tablet), 2times/day(Fasting), take orally, continuous administration until reach the standard of termination.
  Interventions: Drug: Sorafenib Tosylate Tablets

INTERVENTIONS:
Drug: Icaritin — 600mg/time, 6 capsules/time(6×100mg/capsule), 2 times/day(30 minutes after breakfast, lunch and dinner), take orally, continuous administration until reach the standard of termination.
  Arms: Icaritin
Drug: Sorafenib Tosylate Tablets — 400mg/time, 2 tablets/time(2×200mg/tablet), 2times/day(Fasting), take orally, continuous administration until reach the standard of termination.
  Arms: Sorafenib Tosylate Tablets

SUMMARY:
The primary efficacy index of this study is to compare the OS of the two groups.

DETAILED DESCRIPTION:
Icaritin is a newly discovered small molecular compound which is high selective ERa36 modulators ,the preclinical PK&PD and toxicity studies showed it can inhibit the growth of HCC cancer cells both in vitro and in vivo, combining clinical data perhaps it will be a very promising new drug to treat hepatocellular carcinoma (HCC) by targeting this nongenomic pathway. Shenogen decided to further investigate the efficacy and safety of Icaritin and to explore potential gene targets for treating HCC.

The results of phase I study showed Icaritin has good safety and tolerance. The biological availability of Icaritin after meal is high and the half-life is relatively short.

The phase Ib study enrolled 28 subjects. Among the 18 HCC subjects, 12 subjects received treatment in the oral administration group with 600 mg once, twice per day, after meal 30 minutes, 6 subjects received treatment in the oral administration group with 800 mg once, twice per day, after meal 30 minutes. The results showed that in the 600mg group there are 12 HCC patients whose therapeutic efficacy is evaluable now, one case of PR (10%), 5 cases of SD (50%) and 4 cases of PD (40%) were observed.Safety data showed that totally 24 AEs are probably related to investigational drug. Among them, 19 AEs are grade I, 5 AEs are grade II, no grade III or above AE.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet any of the following criteria are not allowed to enter the test:

  1. Aged between 18 and 75 years old, no gender restriction;
  2. According to "Primary Liver Cancer Diagnosis and Treatment Standard." (2011 Edition) issued by the National Health and Family Planning Commission, advanced or metastatic hepatocellular carcinoma patients who diagnosed by pathology /cytology fail to undergo liver surgery and/or other local treatment (ablation or hepatic artery intervention), or have recurrence and progression after surgery and/or other local treatment;
  3. Not previously accepted first-line system therapy (systemic chemotherapy, molecular targeting, immunotherapy and research medication, etc.) for advanced or metastatic HCC, including but not limited to systematic chemotherapy with oxaliplatin, sorafenib, PD-1/PD-L1 antibody and Icaritin, etc.;
  4. The central laboratory must receive specimen of tumor tissue (wax block or white slice) at first, and detect the PD-L1of tumor tissues by immunohistochemistry, only positive expression of PD-L1 in immune cells can be enrolled;
  5. According to the evaluation criteria of solid tumor reaction (RECIST 1.1), it has at least one measurable target lesion (Non-lymph node lesions with the longest diameter larger than 10mm, lymph node lesions with the short diameter larger than 15mm); the lesions previously received local treatment such as ablation or hepatic artery interventional therapy should be detected by computed tomography (CT) / magnetic resonance imaging (MRI) and according to RECIST1.1, It's sure that disease progression has occurred and the longest diameter is more than 1.0cm,it can be used as a measurable target lesions;
  6. Liver surgery was performed more than 3 months ago, ablation or interventional treatment of hepatic artery was performed more than 4 weeks ago, and the adverse reactions returned to normal; After surgery or other local treatment, if patients have gone beyond the norm for systemic adjuvant chemotherapy or sorafenib, it will need more than 6 months after the chemotherapy or sorafenib, and disease progression and / or metastasis have occurred;
  7. The Child-Pugh score of liver function is grade A or better grade B (score≤7);
  8. The ECOG score of physical condition is 0-1;
  9. Expected survival time≥12 weeks;
  10. 2 weeks before the first medication of the trial, there is no use of modern Chinese medicine preparation with liver cancer indication, including Delisheng injection, Kanglaite injection/soft capsule, Aidi injection or Cotside injection, elemene injection/oral liquid, Huaier granule, cinobufotalin and GanFuLe capsule / tablet and so on.
  11. The function of the main organs is basically normal and meets the following requirements:

      ① Marrow: Absolute neutrophil count≥1.5×109/L, platelet≥80×109/L, hemoglobin≥90g/L;

      ② Liver: Total bilirubin≤1.5 times of the upper limit of normal(ULN), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤5 × ULN; albumin≥29g/L;

      ③ Kidney: Serum creatinine≤ 1.5 x ULN, or creatinine clearance rate≥ 50ml/min;
  12. If HBV-DNA≥104 copies/ml(2000IU/ml), antiviral therapy must be done first, the patient can be included in the group until HBV-DNA<104 copies /ml(2000IU/ml); and continue to take antiviral drugs, monitor liver function and hepatitis B virus load;
  13. Women of childbearing age must receive pregnancy tests 14 days before treatment and the results are negative; Men and women must take effective contraceptive measures during the trial (from signing an informed consent to 3 months after the last medication);
  14. Patients volunteered to join the study, sign the informed consent, have good compliance and cooperate with follow-up;
  15. The subjects do not participate in other clinical trials within 4 weeks before screening; If the subject fails in other test screening, but meets the requirements of this test, then can be enrolled.

Exclusion Criteria:

* Patients who meet any of the following criteria are not allowed to enter the test:

  1. Imaging examination shows that HCC liver tumors are huge (≥60% of the liver volume), or cancer embolus of portal trunk (occupying ≥50% of the vascular diameter), or cancer embolus invading mesenteric vein or inferior vena cava;
  2. Middle or higher ascites which is clinically significant, it requires therapeutic abdominal paracentesis /drainage, or the Child-Pugh score > 2;
  3. Local anticancer therapy (including surgery, ablation, hepatic arterial chemotherapy, embolization or radiotherapy) or major surgery was performed 28 days prior to randomization;
  4. Hepatocholangiocarcinoma and fibrolamellar cell carcinoma; In the past or at the same time, there were other cancers whose primary site or histology are entirely different from hepatocellular carcinoma, except cervical carcinoma in situ, previously treated basal cell carcinoma and superficial bladder tumor (Ta, Tis, T1); Patients with other malignancies who have been cured for >5 years prior to enrollment may be admitted to the group;
  5. Pregnant or lactating women;
  6. Patients who have high blood pressure and failed to receive good control with antihypertensive drugs (systolic blood pressure >140mmHg, diastolic pressure >100mmHg); Patients suffer from CTCAE classification type II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmia; and/or New York Heart Association(NYHA) grade III to IV cardiac dysfunction.
  7. Allograft transplants including liver transplantation were performed previously, or a liver transplant was planned during the trial;
  8. Hepatic encephalopathy and / or hepatic nephropathy occurred within 6 months;
  9. Patient with active hepatitis C, that is, anti -HCV positive or HCV-RNA positive and abnormal liver function;
  10. Human immunodeficiency virus (HIV) tests are positive or severe infection requiring systemic treatment with antibiotics;
  11. Inability to swallow, chronic diarrhea or intestinal obstruction that significantly affecting medication intake and absorption;
  12. Having a history of digestive tract bleeding within 6 months, or with a clear gastrointestinal bleeding tendency, including local active ulcerative lesions, positive fecal occult blood;
  13. The patient has or is suspected to have known active autoimmune disease;
  14. If a central nervous system metastasis is known and a metastasis of the central nervous system is suspected, the cranial MRI examination should be performed to exclude it;
  15. Abnormal coagulation function: prothrombin time (PT) >16S or international normalized ratio (INR) >1.5;
  16. There is a history of schizophrenia or psychotropic substance abuse;
  17. Known to be allergic or intolerant to Icaritin or sorafenib and excipients;
  18. Other conditions that researchers believe discourage patients from participating in trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 1-2 years
  OS is defined as the time from randomization to died from any cause. For the subjects who failed to visit, deletion is performed on the final date of knowing the survival of the subjects, for subjects who still survive, deletion is performed on the data expiration date.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1-2 years
  PFS is defined as the date from randomization to the first radiographic record of disease progression or death (whichever occurs first). See the Statistical Analysis Plan (SAP) for the definition of PFS deletion rule.
Time to progress（TTP） | 1-2 years
  TTP is defined as the date from randomization to the first radiographic record of disease progression, see the Statistical Analysis Plan(SAP) for the definition of TTP deletion rule.
Overall response rate (ORR) | 1-2 years
  ORR is defined as the proportion of subjects achieving optimal overall efficacy such as CR or partial remission (PR).
Overall disease control rate (DCR) | 1-2 years
  DCR is defined as the proportion of subjects achieving optimal overall efficacy such as CR, PR or stable disease (SD).
Assessment on Quality of life 1 | 1-2 years
  Quality of life (QOL) changes: Quality of life scores are assessed with EORTC QLQ-C30 and compared with baseline values.
Assessment on Quality of life 2 | 1-2 years
  Quality of life (QOL) changes: Quality of life scores are assessed with EORTCQLQ-HCC-18 and compared with baseline values.

OTHER OUTCOMES:
Biomarker analysis of proteome level (Immunohistochemical method) | 1-2 years
  Baseline expression or expression changes of programmed cell death ligand 1 (PD-L1), heterogeneous ribonucleoprotein A2/B1 (hnRNPAB1) and interleukin -6 (IL-6) and so on.
Genome level (DNA, mRNA, miRNA) biomarker analysis | 1-2 years
  Genetic variation(Liver cancer driver genes and hotspot gene mutations, such as IDH1/2, JAK2/3, PD-L1/2), expression levels of oncogenes and immune related genes(Gene copy number and RNA expression level) and epigenetics cohort analysis

CONTACTS AND LOCATIONS:
Overall Officials: Yan Sun, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Shukui Qin, MD, Principal Investigator — NanJing PLA 81 Hospital
Locations (26):
- China (26):
  - First Affiliated Hospital Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Cancer institute & hospital, chinese academy of medical sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - The fifth medical center of PLA General Hospital, Beijing, Beijing Municipality
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Eastern Theater General Hospital,QinHuai District Medical Area, Nanjing, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - Jilin Cancer Hospital, Changchun, Jilin
  - Jinan Central Hospital, Jinan, Shandong
  - Linyi Tumour Hospital, Linyi, Shandong
  - Fudan University Affiliated Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institution & Hospital, Tianjin, Tianjin Municipality
  - Nanfang Hospital of Southern Medical University, Guangzhou